CLINICAL TRIAL: NCT02000791
Title: Does Laryngoscopic Tecnique Facilitate cLMA Insertion?
Acronym: cLMA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tugba Arslan, medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: laryngeal mask
Record Dates: First submitted 2013-11-21; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Urologic Surgery
Keywords: cLMA; laryngoscopy; fiberoptic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cLMA insertion via laryngoscopic technique (Experimental): Comparison of cLMA insertion via laryngoscope view by fiberscope
  Interventions: Other: Comparison of fibreoptic view
- cLMA insertion via standart technique (Active Comparator): Comparison of cLMA insertion via standart technique view by fiberscope
  Interventions: Other: Comparison of fibreoptic view

INTERVENTIONS:
Other: Comparison of fibreoptic view

SUMMARY:
it is compared that laryngeal mask insertion with standard technique and laryngoscopic technique

DETAILED DESCRIPTION:
Is there any releation between insertion succes rate and difficult intubation criteria. success of the first attempt laryngeal mask insertion, patient response of laryngeal mask placement. And also during the implementation of these two techniques; the effects on heart rate and blood pressure and postoperative complications were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 age
* under urologic surgery patient

Exclusion Criteria:

* Uper respiratory infection
* Full stomach
* BMI over 40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-02 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
İnvestigate to easy of insertion whether standart or laryngoscopic technique | 1 min after insertion

SECONDARY OUTCOMES:
Fiberoptic view | 1 min after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Arslan, MD, Principal Investigator
Locations (1):
- Diskapi Yildiim Beyazit Eduation and Research Hospital, Ankara, Turkey (Türkiye)